CLINICAL TRIAL: NCT02606604
Title: Effects of Functional Electrical Stimulation Cycling Versus Cycling Only on Walking Performance and Quality of Life in Individuals With Multiple Sclerosis: A Pilot Study
Brief Title: Effects of Functional Electrical Stimulation Cycling Versus Cycling Only on Walking and Quality of Life in MS
Acronym: MSCycling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Lori Hochman, Clinical Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 534378-1
Record Dates: First submitted 2015-03-19; First posted 2015-11-17 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Multiple Sclerosis
Keywords: Functional Electrical Stimulation; Cycling
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FES Cycling (Experimental): The intervention consists of electrical stimulation to five lower extremity muscle groups (quadricep, hamstring, anterior tibialis, gluteal, and gastrocnemius muscle groups) while cycling for 45 minutes, 3 times per week for 8 weeks. Outcome measures will be collected at baseline, 4 weeks, 8 weeks and 4 weeks after training is completed).
  Interventions: Device: RT 300: Lower Extremity Cycling
- Cycling Only (Active Comparator): The intervention consists of lower extremity cycling for 45 minutes, 3 times per week for 8 weeks. Electrical stimulation will not be applied to any muscles. Outcome measures will be collected at baseline, 4 weeks, 8 weeks and 4 weeks after training is completed.
  Interventions: Device: RT 300: Lower Extremity Cycling

INTERVENTIONS:
Device: RT 300: Lower Extremity Cycling — Individuals will be randomly assigned to either the FES cycling or cycling only group and will perform lower extremity cycling. Individuals will participate in an interval training cycling program 3 times per week for 8 weeks.
  Other Names: RT 300; Lower Extremity Ergometer

SUMMARY:
This study will seek to determine the benefits that FES-LE cycling has over cycling alone on walking performance and quality of life in people with multiple sclerosis.

DETAILED DESCRIPTION:
Functional Electrical Stimulation (FES) is a rehabilitation tool that stimulates nerves via electrical current, causing muscles to contract. When FES is appled to leg muscles during stationary cycling the legs move in a fixed rhythmical pattern. Previous studies have demonstrated that FES during cycling is a safe and effective exercise for individuals recovering from spinal cord injury or stroke, but few have applied this tool to a progressive disorder, such as multiple sclerosis (MS). The aim of this study is to assess the immediate and short-term effect of an 8-week training program comparing FES lower extremity cycling to cycling without FES. Twenty volunteers with MS will participate. They will be randomly assigned to a training group. This study examine the effects of training on quality of life, endurance, walking speed, and step quality. Participants will sign an informed consent and complete a questionnaire that includes medical history and demographic data. Before training, immediately after training finishes and one month after training, self-report questionnaires, timed walking tests will be completed. During the walking tests, step quality and speed will be measured with a sensor that is worn on a belt

ELIGIBILITY:
Inclusion Criteria:

* Medical Diagnosis of MS
* Patient-determined Disease Steps score between 3.0 and 6.0 inclusive
* Ability to attend training sessions 3 times per week for an 8-10 week period
* Passing a submaximal exercise test
* Adequate hip range of motion (at least 110 degrees)
* Adequate knee range of motion (10-90 degrees)

Exclusion Criteria:

* Cognitive deficits that would interfere in ability to sign consent and understand the procedures for the study.
* History or presence of other neurological pathologies that interfere with movement
* Received physical therapy within the last 4 weeks prior to the study
* History of an acute exacerbation of their MS symptoms within 4 weeks prior to the study
* Immunosuppressive or steroid therapy within the past 4 weeks
* Significant spasticity in the legs that interferes with the cycling motion
* History of congestive heart failure
* Coronary Artery Disease
* Uncontrolled Hypertension
* History of epilepsy or seizures
* Cardiac demand pacemaker or implanted defibrillator
* Unhealed fractures in the legs
* Pressure sores or open wounds on the legs
* Pregnant or trying to conceive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori I Hochman, PT, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook Univeristy, Stony Brook, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PWMS were recruited from various sources from including: physician practices, physical therapy practices, support groups, web postings, email, fitness centers, and personal communication. Recruitment was from June 2015 - July 2017.
Pre-assignment Details: Participants were excluded from the study if they did not meet the inclusion/exclusion criteria.
Groups:
- Functional Electrical Stimulation Cycling: The intervention consisted of electrical stimulation to five lower extremity muscle groups (quadricep, hamstring, anterior tibialis, gluteal, and gastrocnemius muscle groups) while cycling for 45 minutes, 3 times per week for 8 weeks for a total of 24 sessions. Outcome measures were collected at baseline, 4 weeks, 8 weeks and 4 weeks after training was completed. Seven subjects completed this arm of the intervention.
- Cycling Only: The intervention consisted of lower extremity cycling for 45 minutes, 3 times per week for 8 weeks for at total of 24 sessions. Electrical stimulation was not be applied to any muscles. Outcome measures were collected at baseline, 4 weeks, 8 weeks and 4 weeks after training is completed. Seven subjects completed this arm of the intervention.
Period: Overall Study
Arm/Group | Functional Electrical Stimulation Cycling | Cycling Only
Started | 8 | 7
Completed | 7 | 7
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FES Cycling | Cycling Only | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 11
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.71 (7.54) | 47.51 (8.97) | 53.64 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 4 | 2 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 14
Patient Determined Disease Steps (PPDS) [Mean (Standard Deviation); unit: units on a scale] — PPDS is a self-report measure that determines level of disability and disease stage of people with multiple sclerosis. This scale ranges from 0 to 8, with 0 = no disability and 8 = bed-ridden.
  units on a scale | 3.71 (.76) | 3.71 (1.11) | 3.71 (.91)

OUTCOME MEASURES:

1. Primary Outcome: Gait Velocity: Timed Walking
Description: Gait velocity was reported in meters/second based on a 25 foot walk test called the Timed 25 foot Walk Test. Faster gait speeds are better outcomes.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: meters/second
Groups:
- FES Cycling: The intervention consisted of electrical stimulation to five lower extremity muscle groups (quadricep, hamstring, anterior tibialis, gluteal, and gastrocnemius muscle groups) while cycling for 45 minutes, 3 times per week for 8 weeks for a total of 24 sessions. Outcome measures were collected at baseline, 4 weeks, 8 weeks and 4 weeks after training was completed. Seven subjects completed this arm of the intervention. One participant withdrew after the second session of cycling due to developing neck pain and did not continue with the study.
- Cycling Only: The intervention consisted of lower extremity cycling for 45 minutes, 3 times per week for 8 weeks for at total of 24 sessions. Electrical stimulation was not be applied to any muscles. Outcome measures were collected at baseline, 4 weeks, 8 weeks and 4 weeks after training is completed. Eight subjects completed this arm of the intervention.
Arm/Group | FES Cycling | Cycling Only
Number analyzed (Participants) | 7 | 7
meters/second | 1.33 (1.39) | 1.4 (1.48)

2. Primary Outcome: Gait Velocity: Timed Walking
Description: as for outcome 1
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: meters/second
Arm/Group | FES Cycling | Cycling Only
Number analyzed (Participants) | 7 | 7
meters/second | 1.34 (.18) | 1.42 (.18)

3. Primary Outcome: Gait Velocity: Timed Walking
Description: as for outcome 1
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: meters/second
Arm/Group | FES Cycling | Cycling Only
Number analyzed (Participants) | 7 | 7
meters/second | 1.39 (.18) | 1.45 (.18)

4. Primary Outcome: Gait Velocity: Timed Walking
Description: as for outcome 1
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: meters/second
Arm/Group | FES Cycling | Cycling Only
Number analyzed (Participants) | 7 | 7
meters/second | 1.44 (.18) | 1.42 (.18)

5. Secondary Outcome: Self-reported Fatigue Using Modified Fatigue Impact Scale
Description: The Modified Fatigue Impact Scale is a 21 item self-report questionnaire that takes 5-10 minutes to complete. It uses a 5-point likert scale to rate the patient's perception of how Multiple Sclerosis related fatigue affects an individual's life on an everyday basis. It contains three subscales that include: cognitive, physical, and psychosocial dimensions. Scores on the subscales can be analyzed individually or as a summed score to give an overall fatigue score. Higher scores indicate a greater impact of fatigue. The minimum score is a 0 and the maximum score is 81.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FES Cycling | Cycling Only
Number analyzed (Participants) | 7 | 7
score on a scale | 42 (6.19) | 47.13 (6.19)

6. Secondary Outcome: Self-reported Fatigue Using Modified Fatigue Impact Scale
Description: as for outcome 5
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FES Cycling | Cycling Only
Number analyzed (Participants) | 7 | 7
score on a scale | 32 (6.19) | 39.57 (6.19)

7. Secondary Outcome: Self-reported Walking Using 12 Item Multiple Sclerosis Walking Scale
Description: The Multiple Sclerosis Walking Scale is a 12-item self-report questionnaire that takes approximately 10 minutes to complete and reflects a persons' perception of the impact that multiple sclerosis has on walking ability during the past 2 weeks. Each of the items scored ranges from 1 to 5, in which higher scores indicate a greater impact of multiple sclerosis on their walking. Scores on the 12 items are summed. To transform to a 0-100 scale, the minimum score of 12 is subtracted from the sum; the result is divided by 48 and then multiplied by 100. The lowest score is 0 and the highest score is 100. Higher scores mean a worse outcome.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FES Cycling | Cycling Only
Number analyzed (Participants) | 7 | 7
score on a scale | 64.43 (6.78) | 71.43 (6.78)

8. Secondary Outcome: Self-reported Walking Using 12 Item Multiple Sclerosis Walking Scale
Description: as for outcome 7
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FES Cycling | Cycling Only
Number analyzed (Participants) | 7 | 7
score on a scale | 59.91 (6.68) | 69.52 (6.78)

9. Secondary Outcome: Overall Self-reported Quality of Life Using Multiple Sclerosis Quality of Life- 54
Description: The Multiple Sclerosis Quality of Life-54 is a self-report quality of life questionnaire. It measures health-related quality of life using both generic and disease-specific measures and was constructed by experts in the field. There is no overall score for this scale since it contains 12 subscales, two summary scores, and two single-item measures. The quality of life subscale was the chosen outcome measure reported below. The scores range from 0-100. Higher scores on the scale notes improved outcome.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FES Cycling | Cycling Only
Number analyzed (Participants) | 7 | 7
score on a scale | 61.19 (6.28) | 57.62 (6.28)

10. Secondary Outcome: Overall Self-reported Quality of Life Using Multiple Sclerosis Quality of Life- 54
Description: as for outcome 9
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FES Cycling | Cycling Only
Number analyzed (Participants) | 7 | 7
score on a scale | 70.95 (6.28) | 60.95 (6.28)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks.
Arm/Group | FES Cycling | Cycling Only
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT02606604/Prot_SAP_000.pdf